CLINICAL TRIAL: NCT04646785
Title: Mindfulness-based Cognitive Therapy to Improve Stress and Sleep in Patients With Inflammatory Bowel Disease
Brief Title: Mindfulness-based Cognitive Therapy for Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Jeroen Bosch Ziekenhuis (Other); Rijnstate Hospital (Other); Canisius-Wilhelmina Hospital (Other); Donders Centre for Cognitive Neuroimaging (Other)
Responsible Party: Principal Investigator, Anne Speckens, Principal Investigator and Director of Radboudumc Centre for Mindfulness, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MBCT-IBD-2020-2024
Record Dates: First submitted 2020-11-16; First posted 2020-11-30 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: randomized controlled trial; mindfulness-based cognitive therapy; effectiveness; psychological distress; sleep; fatigue
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fatigue | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: A randomized, multicenter, clinical trial with assessments at baseline, post treatment (3 months later) and follow-ups at 6, 9 and 12 months after baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based cognitive therapy (MBCT) added to treatment as usual (Experimental): Patients in the MBCT arm will in addition to their treatment as usual be invited to participate in MBCT.
  Interventions: Behavioral: Mindfulness-based cognitive therapy + TAU
- Treatment as usual (TAU) (Active Comparator): Patients in this arm will receive treatment as usual.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy + TAU — The proposed intervention is mindfulness-based cognitive therapy (MBCT), based on the protocol published by Segal, Williams and Teasdale. MBCT consists of eight weekly 2.5h group sessions, a six-hour silent day and daily home practice assignments guided by audio files. The program includes both formal and informal meditation exercises. Cognitive techniques include monitoring and scheduling of activities, identification of negative automatic thoughts and devising a relapse prevention plan. Psycho-education and interactive dialogue typically focus on stress management, balancing activities, and (lifestyle) strategies to stay well in the future (relapse prevention).
  Arms: Mindfulness-based cognitive therapy (MBCT) added to treatment as usual
Other: Treatment as usual (TAU) — Treatment as usual (TAU) according Dutch and European IBD treatment guidelines. TAU focuses on pharmacological and surgical disease control, and prevention of complications.
  Arms: Treatment as usual (TAU)

SUMMARY:
Considering the limited availability of psychosocial interventions for IBD, this study aims to investigate MBCT as an adjunctive treatment to treatment as usual to reduce psychological stress and improve sleep quality/regularity in patients with IBD who report elevated stress levels. The study will have a follow-up duration of 12 months from baseline.

DETAILED DESCRIPTION:
Introduction:

Inflammatory bowel diseases (IBD) are chronic inflammatory diseases of the intestinal tract, consisting of crohn's disease (CD) and ulcerative colitis (UC). In The Netherlands, there are about 90,000 IBD patients, mainly young adults who are in a turbulent part of their life with starting a family and career. The prevalence of IBD seems to be rising. The peak incidence is between 15 and 30 years. The disease is characterized by periods of disease activity (flares) alternating with periods of (clinical) remission. Physical symptoms include abdominal pain, diarrhea, rectal bleeding and fatigue. Although the arsenal of drugs has increased in recent decades, there is no cure for the disease and patients are usually long-term treated with different (immunosuppressive) medications. Nevertheless, at this moment, we are only partially able to keep our IBD patients in remission.

Even in those in remission, IBD is associated with increased levels of psychological stress, with estimated prevalence rates of 21% for depressive symptoms and 35% for anxiety symptoms. In periods of disease activity, prevalence of elevated anxiety levels was even found to be as high as 75.6%. Besides psychological stress, IBD patients in remission report lower quality of life compared to the general population. This is due to the physical symptoms but also to fatigue, worries, anxiety, depression, impaired satisfaction with social role and sleep disturbances. More than 40 % of the IBD patients experience fatigue. This may contribute to the higher sick leave days and higher work impairment rates in quiescent IBD, causing high societal costs. In addition, poor sleep seems common in individuals with IBD and has been linked to disease activity and shown as a predictor for subclinical inflammation and a risk factor for relapse and poorer outcomes.

Mindfulness training, typically in the form of mindfulness-based stress reduction (MBSR) or mindfulness-based cognitive therapy (MBCT), is a psychosocial group-based intervention that has been shown to reduce psychological distress and improving quality of life, both in patients with mental health problems and those with chronic diseases such as diabetes, cancer, cardiovascular disease, rheumatoid arthritis and fibromyalgia. Mindfulness training focuses on the progressive acquisition of mindful awareness to better cope with negative repetitive thoughts and feelings, and for that reason may be a good option to reduce psychological stress and fatigue, and improve quality of life in patients with chronic conditions including IBD.

Although the available literature on the effectiveness of mindfulness-based interventions for IBD is still relatively scarce, a recent meta-analysis showed significant benefits in terms of stress, depression, and quality of life. However, the variety in types of interventions was rather high, and individual studies typically suffered from methodological limitations, including small sample size, poor blinding of the outcome assessors, incomplete data reporting and a relative lack of fidelity measures. Therefore, it seems warranted to conduct a high-quality, multicenter randomized controlled trial investigating the effectiveness of MBCT to improve stress, sleep quality, and quality of life.

Aims:

Considering the limited availability of psychosocial interventions for IBD, this study aims to investigate MBCT as an adjunctive treatment to TAU to reduce psychological stress in patients with IBD who report elevated stress levels. In addition, we aim to improve sleep quality/regularity and fatigue, IBD-related quality of life, perceived control over IBD, clinical indicators (fecal calprotectin, c-reactive protein levels, Harvey Brashaw Index for CD, Simple Clinical Colitis Activity Index for UC), IBD-related flare. We also aim to improve repetitive negative thinking, mindfulness skills, self-compassion skills, and positive mental health. We will investigate whether improving sleep quality may be one of the pathways through which mindfulness may help reduce psychological distress and improve quality of life in IBD (working mechanism).

Method:

A two-armed randomized, multicenter, parallel group pragmatic trial comparing Mindfulness-Based Cognitive Therapy (MBCT) vs. Treatment As Usual (TAU) for reducing psychological distress in distressed patients with Inflammatory Bowel Disease (IBD). Assessments will be conducted at baseline, post treatment (3 months) and follow-ups at 6, 9, and 12 months. Objective sleep measures will be taken at baseline, post treatment and 12 months.

The control group will receive treatment as usual (TAU) according to Dutch and European IBD treatment guidelines. The intervention group will receive Mindfulness-Based Cognitive Therapy (MBCT) in addition to TAU. The MBCT protocol that will be used is based on the protocol published by Segal, Williams and Teasdale. MBCT consists of eight weekly 2.5h group sessions, a six-hour silent day and daily home practice assignments guided by audio files. Mindfulness is characterized by deliberate, non-judging and sustained moment-to-moment awareness. Health related benefits include enhanced emotional processing and coping regarding the effects of chronic illness and stress, improved self-efficacy and control, and a more accepting attitude towards difficult emotions, thought and bodily sensations. Psycho-education and interactive dialogue typically focus on stress management, balancing activities, lifestyle factors, and strategies to stay well in the future (relapse prevention). Each group will be comprising 8-12 participants. MBCT courses will be taught on site by qualified mindfulness teachers. Teacher competency will be assessed with the Mindfulness-Based Interventions - Teaching Assessment Criteria, using a random selection of videotaped sessions, assessed by expert teachers who have been trained to use these assessment criteria.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed IBD diagnosis of Crohn's disease (CD), Ulcerative colitis (UC) or Indeterminate colitis (IC)
* Current IBD remission (Calprotectin < 250 mg/kg) since at least three months
* Hospital Anxiety and Depression Scale-score of >=11, indicating at least mild levels of psychological distress (Vodermaier 2011).
* Age of 16 or older
* Taking no IBD medication or on a stable dose of 5-ASA products, immunosuppressive medication, or biologics for at least three months prior to enrollment.

Exclusion Criteria:

* Severe psychiatric disorders (e.g. acute suicidality, psychosis)
* Current alcohol or drug dependency
* Untreated anemia
* Prior participation in an 8-week MBSR or MBCT-programme

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Psychological distress | Change between baseline and 3 months
  Measured by the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items, 7 related to depression and 7 related to anxiety. Scoring for each item ranges from zero to three. Three denotes highest anxiety or depression level meaning that a person can score between 0 and 21 for either anxiety or depression.
Psychological distress | Change between 3 and 12 months
  Measured by the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items, 7 related to depression and 7 related to anxiety. Scoring for each item ranges from zero to three. Three denotes highest anxiety or depression level meaning that a person can score between 0 and 21 for either anxiety or depression.

SECONDARY OUTCOMES:
Objective sleep quality | Change between baseline and 3 months
  operationalized as total sleep time, time spent in slow wave sleep, sleep continuity, all measured with wearable sleep EEG (iBand+/ Arenar and Fitbit activity tracker).
Objective sleep quality | Change between 3 and 12 months
  operationalized as total sleep time, time spent in slow wave sleep, sleep continuity, all measured with wearable sleep EEG (iBand+/ Arenar and Fitbit activity tracker).
Subjective sleep quality | Change between baseline and 3 months
  Measured by the Pittsburgh Sleep Quality Inventory (PSQI). The PSQI consist of 19 items offering 7 components scores and one composite score. Scoring for each component ranges from zero to three. The overall PSQI score is then calculated by totaling the seven component scores, providing an global score ranging from zero to twenty-one. Lower scores indicate a healthier sleep quality.
Subjective sleep quality | Change between 3 and 12 months
  Measured by the Pittsburgh Sleep Quality Inventory (PSQI). The PSQI consist of 19 items offering 7 components scores and one composite score. Scoring for each component ranges from zero to three. The overall PSQI score is then calculated by totaling the seven component scores, providing an global score ranging from zero to twenty-one. Lower scores indicate a healthier sleep quality.
Fatigue | Change between baseline and 3 months
  measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F).The FACIT-F is a 40-item self-reported measure that assesses fatigue and its impact on daily activities and function. Subdomains include: physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being and Fatigue. The subdomain fatigue consists of 13-items. Items are scored on a 0-4 response scale with anchors ranging from 'not at all' to 'very much so'. All items are summed to create a global fatigue score with a range from 0 to 52. Higher scores indicate increased fatigue.
Fatigue | Change between 3 and 12 months
  measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F).
IBD-related quality of life | Change between baseline and 3 months
  measured by the Inflammatory Bowel Disease Quality of Life Questionnaire (IBDQ). The IBDQ has 32 items scored on a 7-point Likert scale, ranging from 1 (worst health) to 7 (best health). Overall score range from 32 to 224, with higher scores reflecting better quality of life.
IBD-related quality of life | Change between 3 and 12 months
  measured by the Inflammatory Bowel Disease Quality of Life Questionnaire (IBDQ). The IBDQ has 32 items scored on a 7-point Likert scale, ranging from 1 (worst health) to 7 (best health). Overall score range from 32 to 224, with higher scores reflecting better quality of life.
Perceived control over IBD | Change between baseline and 3 months
  measured by the IBD-Control questionnaire. The IBD-Control Questionnaire consists of eight items, which generate an overall score ranging from 0 (worst control) to 16 (best control).
Perceived control over IBD | Change between 3 and 12 months
  Measured by the IBD-Control questionnaire. The IBD-Control Questionnaire consists of eight items, which generate an overall score ranging from 0 (worst control) to 16 (best control).
Calprotectin | Change between baseline and 3 months
  Assessed in accordance with regular medical procedures. Having higher levels of calprotectin generally means that there is active inflammation in the body or intestines. For a calprotectin test, a normal reading is less than 100 mcg/g.
Calprotectin | Change between 3 and 12 months
  Assessed in accordance with regular medical procedures. Having higher levels of calprotectin generally means that there is active inflammation in the body or intestines. For a calprotectin test, a normal reading is less than 100 mcg/g.
C-reactive protein levels | Change between baseline and 3 months
  Assessed in accordance with regular medical procedures. Also having higher levels of c-reactive protein generally means that there is active inflammation in the body or intestines. For a CRP test, a normal reading is less than 10 milligram per liter (mg/L).
C-reactive protein levels | Change between 3 and 12 months
  Assessed in accordance with regular medical procedures. Also having higher levels of c-reactive protein generally means that there is active inflammation in the body or intestines. For a CRP test, a normal reading is less than 10 milligram per liter (mg/L).
Clinical disease activity | change between baseline and 3 months
  Assessed by a clinician with the Harvey Brashaw Index (HBI) for Crohn's disease and the Simple Clinical Colitis Activity Index
Clinical disease activity | change between 3 and 12 months
  Assessed by a clinician with the Harvey Brashaw Index (HBI) for Crohn's disease and the Simple Clinical Colitis Activity Index
Repetitive negative thinking | Change between baseline and 3 months
  measured by the 15-item Perseverative Thinking Questionnaire (PTQ). The PTQ is a 15-item self-report questionnaire. Respondents are asked to describe how they typically think about negative experiences or problems. They rate each item on a 5-point Likert scale from 0 (never) to 4 (almost always) the extent to which each statement applies to them when they think about negative experiences or problems. All items are summed to create a global repetitive negative thinking score ranging from 0 to 60. Higher scores indicate increased repetitive negative thinking.
Repetitive negative thinking | Change between 3 and 12 months
  measured by the 15-item Perseverative Thinking Questionnaire (PTQ). The PTQ is a 15-item self-report questionnaire. Respondents are asked to describe how they typically think about negative experiences or problems. They rate each item on a 5-point Likert scale from 0 (never) to 4 (almost always) the extent to which each statement applies to them when they think about negative experiences or problems. All items are summed to create a global repetitive negative thinking score ranging from 0 to 60. Higher scores indicate increased repetitive negative thinking.
Mindfulness skills | Change between baseline and 3 months
  24-item Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF). This questionnaire is divided into the subscales observing, describing, acting with awareness, non-judging and non-reactivity.
Mindfulness skills | Change between 3 and 12 months
  24-item Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF). This questionnaire is divided into the subscales observing, describing, acting with awareness, non-judging and non-reactivity.
Positive mental health | Change between baseline and 3 months
  Measured by the Mental Health Continuum-Short Form (MHC-SF). MHC-SF consists of 14-items and assesses emotional, psychological and social well-being. All items are summed and then a mean score is calculated, which represents a global positive mental health score ranging from 0 to 5. Higher scores indicate a better positive mental health.
Positive mental health | Change between 3 and 12 months
  Measured by the Mental Health Continuum-Short Form (MHC-SF). MHC-SF consists of 14-items and assesses emotional, psychological and social well-being. All items are summed and then a mean score is calculated, which represents a global positive mental health score ranging from 0 to 5. Higher scores indicate a better positive mental health.
Self-compassion | Change between baseline and 3 months
  We will use the 12-item Dutch short-form version of the SCS-SF to measure self-compassion. The scale consists of six components, including self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. In the short form, each scale consists of 2 items scored between 1 ((almost) never) to 7 ((almost) always) and subscale score ranges between 2 and 14. A higher score indicates a higher level of self-kindness, common humanity, and mindfulness, and lower scores of self-judgment, isolation, and over-identification. Total scores range from 12 to 84 (summed subscale scores), a higher score indicates a higher level of self-compassion.
Self-compassion | Change between 3 and 12 months
  We will use the 12-item Dutch short-form version of the SCS-SF to measure self-compassion. The scale consists of six components, including self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. In the short form, each scale consists of 2 items scored between 1 ((almost) never) to 7 ((almost) always) and subscale score ranges between 2 and 14. A higher score indicates a higher level of self-kindness, common humanity, and mindfulness, and lower scores of self-judgment, isolation, and over-identification. Total scores range from 12 to 84 (summed subscale scores), a higher score indicates a higher level of self-compassion.
Costs | 12 months
  This will be investigated by using the Trimbos iMTA Questionnaire for Costs associated with Psychiatric Illness (TiC-P) as a measure of healthcare utilization. Unit cost estimates are derived from the national manual for cost prices in the healthcare sector.
Health-related quality of life | 12 months
  This will be assessed by using the EuroQol-5D (EQ-5D-5L). The EQ-5D-5L consist of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This short self-report instrument is used to assess quality adjusted life years.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Speckens, Dr., Principal Investigator — Radboud University Medical Center; Loes Nissen, Dr., Study Chair — Jeroen Bosch Ziekenhuis; Marloes Huijbers, Dr., Study Chair — Radboud University Medical Center
Locations (4):
- Netherlands (4):
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Ziekenhuis, Arnhem
  - Canisius Wilhelmina Ziekenhuis, Nijmegen

IPD SHARING:
Plan to Share IPD: Yes
The authors intend to make the data available to other researchers after completion of the study and will comply with open access procedures, including open access publishing, as much as possible.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: we expect the final report of the primary endpoint of the study December 2024, and we will have an embargo period of 6 months after publication.
Access Criteria: We will use restricted access, such that interested researchers are welcome to contact us with requests for data. The project team will review the quality of the request and grant permission if the request is in accordance with the terms of use drafted by the Radboudumc.
URL: https://www.lcrdm.nl/

REFERENCES:
- [Background] Ewais T, Begun J, Kenny M, Rickett K, Hay K, Ajilchi B, Kisely S. A systematic review and meta-analysis of mindfulness based interventions and yoga in inflammatory bowel disease. J Psychosom Res. 2019 Jan;116:44-53. doi: 10.1016/j.jpsychores.2018.11.010. Epub 2018 Nov 14. PMID 30654993
- [Background] Neuendorf R, Harding A, Stello N, Hanes D, Wahbeh H. Depression and anxiety in patients with Inflammatory Bowel Disease: A systematic review. J Psychosom Res. 2016 Aug;87:70-80. doi: 10.1016/j.jpsychores.2016.06.001. Epub 2016 Jun 6. PMID 27411754
- [Background] Knowles SR, Graff LA, Wilding H, Hewitt C, Keefer L, Mikocka-Walus A. Quality of Life in Inflammatory Bowel Disease: A Systematic Review and Meta-analyses-Part I. Inflamm Bowel Dis. 2018 Mar 19;24(4):742-751. doi: 10.1093/ibd/izx100. PMID 29562277
- [Background] IsHak WW, Pan D, Steiner AJ, Feldman E, Mann A, Mirocha J, Danovitch I, Melmed GY. Patient-Reported Outcomes of Quality of Life, Functioning, and GI/Psychiatric Symptom Severity in Patients with Inflammatory Bowel Disease (IBD). Inflamm Bowel Dis. 2017 May;23(5):798-803. doi: 10.1097/MIB.0000000000001060. PMID 28301432
- [Background] Chavarria C, Casanova MJ, Chaparro M, Barreiro-de Acosta M, Ezquiaga E, Bujanda L, Rivero M, Arguelles-Arias F, Martin-Arranz MD, Martinez-Montiel MP, Valls M, Ferreiro-Iglesias R, Llao J, Moraleja-Yudego I, Casellas F, Antolin-Melero B, Cortes X, Plaza R, Pineda JR, Navarro-Llavat M, Garcia-Lopez S, Robledo-Andres P, Marin-Jimenez I, Garcia-Sanchez V, Merino O, Algaba A, Arribas-Lopez MR, Banales JM, Castro B, Castro-Laria L, Honrubia R, Almela P, Gisbert JP. Prevalence and Factors Associated With Fatigue in Patients With Inflammatory Bowel Disease: A Multicentre Study. J Crohns Colitis. 2019 Aug 14;13(8):996-1002. doi: 10.1093/ecco-jcc/jjz024. PMID 30721954
- [Background] van der Valk ME, Mangen MJ, Leenders M, Dijkstra G, van Bodegraven AA, Fidder HH, de Jong DJ, Pierik M, van der Woude CJ, Romberg-Camps MJ, Clemens CH, Jansen JM, Mahmmod N, van de Meeberg PC, van der Meulen-de Jong AE, Ponsioen CY, Bolwerk CJ, Vermeijden JR, Siersema PD, van Oijen MG, Oldenburg B; COIN study group and the Dutch Initiative on Crohn and Colitis. Healthcare costs of inflammatory bowel disease have shifted from hospitalisation and surgery towards anti-TNFalpha therapy: results from the COIN study. Gut. 2014 Jan;63(1):72-9. doi: 10.1136/gutjnl-2012-303376. Epub 2012 Nov 7. PMID 23135759
- [Background] Burisch J, Jess T, Martinato M, Lakatos PL; ECCO -EpiCom. The burden of inflammatory bowel disease in Europe. J Crohns Colitis. 2013 May;7(4):322-37. doi: 10.1016/j.crohns.2013.01.010. Epub 2013 Feb 8. PMID 23395397
- [Background] Qazi T, Farraye FA. Sleep and Inflammatory Bowel Disease: An Important Bi-Directional Relationship. Inflamm Bowel Dis. 2019 Apr 11;25(5):843-852. doi: 10.1093/ibd/izy334. PMID 30388243
- [Background] Segal, Z. V., Williams, J. M. G., & Teasdale, J. D. (2013). Mindfulness-based cognitive therapy for depression (second).
- [Background] Guo J, Wang H, Luo J, Guo Y, Xie Y, Lei B, Wiley J, Whittemore R. Factors influencing the effect of mindfulness-based interventions on diabetes distress: a meta-analysis. BMJ Open Diabetes Res Care. 2019 Dec 11;7(1):e000757. doi: 10.1136/bmjdrc-2019-000757. eCollection 2019. PMID 31908794
- [Background] Cillessen L, Johannsen M, Speckens AEM, Zachariae R. Mindfulness-based interventions for psychological and physical health outcomes in cancer patients and survivors: A systematic review and meta-analysis of randomized controlled trials. Psychooncology. 2019 Dec;28(12):2257-2269. doi: 10.1002/pon.5214. Epub 2019 Sep 11. PMID 31464026
- [Background] Scott-Sheldon LAJ, Gathright EC, Donahue ML, Balletto B, Feulner MM, DeCosta J, Cruess DG, Wing RR, Carey MP, Salmoirago-Blotcher E. Mindfulness-Based Interventions for Adults with Cardiovascular Disease: A Systematic Review and Meta-Analysis. Ann Behav Med. 2020 Jan 1;54(1):67-73. doi: 10.1093/abm/kaz020. PMID 31167026
- [Background] Zhou B, Wang G, Hong Y, Xu S, Wang J, Yu H, Liu Y, Yu L. Mindfulness interventions for rheumatoid arthritis: A systematic review and meta-analysis. Complement Ther Clin Pract. 2020 May;39:101088. doi: 10.1016/j.ctcp.2020.101088. Epub 2020 Jan 11. PMID 31957665
- [Background] Haugmark T, Hagen KB, Smedslund G, Zangi HA. Mindfulness- and acceptance-based interventions for patients with fibromyalgia - A systematic review and meta-analyses. PLoS One. 2019 Sep 3;14(9):e0221897. doi: 10.1371/journal.pone.0221897. eCollection 2019. PMID 31479478
- [Background] Crane RS, Eames C, Kuyken W, Hastings RP, Williams JM, Bartley T, Evans A, Silverton S, Soulsby JG, Surawy C. Development and validation of the mindfulness-based interventions - teaching assessment criteria (MBI:TAC). Assessment. 2013 Dec;20(6):681-8. doi: 10.1177/1073191113490790. Epub 2013 Jun 21. PMID 23794181
- [Derived] Ter Avest MM, Huijbers MJ, Horjus CS, Romkens TEH, Witteman EM, van Dop WA, Dresler M, Donders ART, Dijkstra G, Nissen LHC, Speckens AEM. Group-Delivered Mindfulness-Based Cognitive Therapy to Reduce Psychological Distress and Improve Sleep in Patients With Inflammatory Bowel Diseases: A Multicenter Randomized Controlled Trial (MindIBD). Inflamm Bowel Dis. 2025 Nov 1;31(11):3021-3032. doi: 10.1093/ibd/izaf116. PMID 40658641
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Ter Avest MM, van Velthoven ASM, Speckens AEM, Dijkstra G, Dresler M, Horjus CS, Romkens TEH, Witteman EM, van Dop WA, Bredero QM, Nissen LHC, Huijbers MJ. Effectiveness of Mindfulness-Based Cognitive Therapy in reducing psychological distress and improving sleep in patients with Inflammatory Bowel Disease: study protocol for a multicentre randomised controlled trial (MindIBD). BMC Psychol. 2023 Jun 19;11(1):183. doi: 10.1186/s40359-023-01127-0. PMID 37337261